CLINICAL TRIAL: NCT00428649
Title: Optimization of Selenoprotein P in Chinese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, RBurk, M.D., Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DK58763-opt; R01DK058763 (NIH)
Record Dates: First submitted 2007-01-25; First posted 2007-01-30 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Selenium Deficiency
Keywords: Selenium supplements; Selenoprotein P; Optimization
MeSH Terms: interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (7):
- 1 (Experimental): 20 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 20 µg selenium
- 2 (Experimental): 40 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 40 µg selenium
- 3 (Experimental): 60 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 60 µg selenium
- 4 (Experimental): 80 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 80 µg selenium
- 5 (Experimental): 100 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 100 µg selenium
- 6 (Experimental): 120 µg selenium as selenomethionine
  Interventions: Dietary Supplement: 120 µg selenium
- 7 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: 20 µg selenium — 20 µg selenium as selenomethionine
  Arms: 1
Dietary Supplement: 40 µg selenium — 40 µg selenium as selenomethionine
  Arms: 2
Dietary Supplement: 60 µg selenium — 60 µg selenium as selenomethionine
  Arms: 3
Dietary Supplement: 80 µg selenium — 80 µg selenium as selenomethionine
  Arms: 4
Dietary Supplement: 100 µg selenium — 100 µg selenium as selenomethionine
  Arms: 5
Dietary Supplement: 120 µg selenium — 120 µg selenium as selenomethionine
  Arms: 6
Dietary Supplement: placebo — placebo
  Arms: 7

SUMMARY:
The purpose of this study is to determine the amount of selenium as selenomethionine that is required to optimize selenoprotein P in selenium-deficient Chinese subjects

DETAILED DESCRIPTION:
Selenium is an essential nutrient. The Recommended Dietary Allowance (RDA) for selenium is considered to be the amount required to optimize plasma selenoproteins. There are two selenoproteins present in the plasma: selenoprotein P (Se-P) and glutathione peroxidase 3 (GPX-3). Although the amount of selenium required to optimize GPX-3 has been determined, the amount required to optimize Se-P in the plasma remains unknown. We aim to determine this amount by supplementing selenium deficient subjects with varying amounts of selenium as selenomethionine.

The study will take place in Mianning County, China, where selenium status is low. Approximately 150 people will be screened for eligibility to participate in this study. 98 subjects will be enrolled. Background information obtained from each participant will be: age, height, weight and smoking status.

Subjects will be randomized to a selenium supplement group. The selenium supplement will contain either 0, 20, 40, 60, 80, 100, or 120 µg of selenium as selenomethionine. A CDC worker will visit each participant daily to give them their selenium supplement. The CDC worker will watch them take their supplement and will ask if they have any unanticipated problems. Blood samples of 20 ml will be obtained at weeks 0, 4, 8, 12, 16, 20, 24, 32, and 40. Hair samples and 24-hr urine collections will be obtained at 0, 20 and 40 weeks. The total study duration is 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 17 years or older
* healthy
* resident of Mianning County for at least 1 year
* hematocrit (PCV) of 30 or greater

Exclusion Criteria:

* subject has taken selenium supplements within the year prior to study
* subject plans to relocate during study

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Plasma selenoprotein P levels at 0, 4, 8, 12, 16, 20, 24, 32, and 40 weeks | 40 weeks

SECONDARY OUTCOMES:
Total plasma selenium concentrations at 0, 4, 8, 12, 16, 20, 24, 32, and 40 weeks | 40 weeks
Plasma glutathione peroxidase activity at 0, 4, 8, 12, 16, 20, 24, 32, and 40 weeks | 40 weeks
24hr urinary selenium excretion at 0, 20 and 40 weeks | 40 weeks
Hair selenium levels at 0, 20 and 40 weeks | 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raymond F Burk, M.D., Principal Investigator — Vanderbilt University; Yiming Xia, Ph.D., Study Director — Sichuan CDC, Chengdu
Locations (1):
- Sichuan Center for Disease Control and Prevention (Sichuan CDC), Chengdu, Sichuan, China

REFERENCES:
- [Background] Xia Y, Hill KE, Byrne DW, Xu J, Burk RF. Effectiveness of selenium supplements in a low-selenium area of China. Am J Clin Nutr. 2005 Apr;81(4):829-34. doi: 10.1093/ajcn/81.4.829. PMID 15817859
- [Background] Casey CE, Guthrie BE, Friend GM, Robinson MF. Selenium in human tissues from New Zealand. Arch Environ Health. 1982 May-Jun;37(3):133-5. doi: 10.1080/00039896.1982.10667551. PMID 7092329
- [Derived] Xia Y, Hill KE, Li P, Xu J, Zhou D, Motley AK, Wang L, Byrne DW, Burk RF. Optimization of selenoprotein P and other plasma selenium biomarkers for the assessment of the selenium nutritional requirement: a placebo-controlled, double-blind study of selenomethionine supplementation in selenium-deficient Chinese subjects. Am J Clin Nutr. 2010 Sep;92(3):525-31. doi: 10.3945/ajcn.2010.29642. Epub 2010 Jun 23. PMID 20573787